CLINICAL TRIAL: NCT03799029
Title: Effects of a Cognitive Training Program With Game Elements and a Reward Feedback System on Children, Adolescents and Adults Presenting ADHD: an Experimental Study. A Multi-centred Study: Neuchatel, Fribourg and Lausanne
Brief Title: Effects of a Cognitive Training Program With Game Elements Among ADHD
Acronym: CogtrainADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Fribourg (Other)
Collaborators: Paris West University Nanterre La Défense (Other)
Responsible Party: Principal Investigator, Amelie Dentz, principal investigator Ph.D, University of Fribourg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Fribourg
Record Dates: First submitted 2018-05-28; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: ADHD
Keywords: Cognitive training; treatment; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: will compare the ADHD group with a control group including healthy participants .The experimental study uses a pseudo-randomized, double-blind, controlled multi-center design.Participants will be assigned to an experimental group (cognitive training ) or in a control active group.
Who Masked: Participant, Investigator
Masking Description: Participant are blind on their group assignation. Investigator are blind on group assignation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active control group low-intensity (Active Comparator): Low intensity version of the same cognitive training program Exercice are realized at home using a computer 25 sessions of 30-45 minutes are realized five days per week during 5 weeks
  Interventions: Other: Cognitive training
- experimental training group cognitive training (Experimental): a multifactorial cognitive program that tackles working memory, attention, inhibition, planification and reasoning Exercice are realized at home using a computer 25 sessions of 30-45 minutes are realized five days per week during 5 weeks
  Interventions: Other: Cognitive training
- control healthy participants (No Intervention): Just a control group including healthy participants No intervention

INTERVENTIONS:
Other: Cognitive training — Participants will train at home during 25 sessions (about 45 minutes each) over a maximum of 5 weeks. Investigators will verify compliance via Internet and call participants and their legal guardians once a week. A reward system will be established with participants. Five sessions of metacognition (1 hour each) are added.
  Arms: active control group low-intensity; experimental training group cognitive training

SUMMARY:
This study examines the impact of cognitive training among participants with ADHD in Switzerland

DETAILED DESCRIPTION:
The main aim of the experimental study is to investigate cognitive functioning, behavioral and neural levels in ADHD, both before and after cognitive training where there has been the addition of motivation elements. Near and far transfers effects of this new program are evaluated. For far transfers, ambulatory assessment is used to improve ecological validity. Neural activity has rarely been examined in cognitive training with ADHD participants, and that is why this study also includes FMRI measures. Long-term effects, defined as three and six months following the completion of cognitive training, are also investigated. This study focuses on children, adolescents and adults with ADHD. Indeed, cognitive training effects have been rarely studied over the lifespan.

ELIGIBILITY:
Inclusion Criteria:

-

Participants fulfilling all of the following inclusion criteria are eligible for the study for the patients'group:

1. Age between 6 and 65 years' old
2. ADHD diagnostic by a specialist
3. IQ-score higher than 80 for adult according to (WAIS-IV; Wechsler, 2008) and for children and adolescents according to (WISC-IV; Wechsler, 2003)
4. Treatment with or without medication for ADHD
5. Computer and Internet connexion at home
6. Informed consent from participants and the legal guardian of the minors (under 14 years old) involved - as documented by signature (Appendix Informed Consent Form).

Participants fulfilling all of the following inclusion criteria are eligible for the study for the control group of healthy participants:

1. Age between 6 and 65 years' old
2. No ADHD diagnostic by a specialist
3. IQ-score higher than 80 for adult according to (WAIS-IV; Wechsler, 2008) and for children and adolescents according to (WISC-IV; Wechsler, 2003)
4. No medication treatment for ADHD
5. Informed consent from participants and the legal guardian of the minors involved - as documented by signature (Appendix Informed Consent Form).

Exclusion Criteria:

* Exclusion criteria

The exclusion criteria for the participants in the patient's group are:

1. Age younger than 6 and older than 65 years' old
2. No diagnosis of ADHD
3. IQ-score lower than 80 points according to (WAIS-IV; Wechsler, 2008) and for children and adolescents according to (WISC-IV; Wechsler, 2003)
4. No computer and Internet access at home
5. No written consent from participants and from the legal guardians of minors involved as less than 14 years old.

(7) FMRI exclusion: claustrophobia, Pregnancy known or suspected,metallic implants in their bodies (e.g: pacemakers, aneurism clips, metal Prosthetic, cochlear implant) (8) In case of suicidal risk, the participant is encouraged to consult the medical staff (9) Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant (10) Participation in another study on cognitive training (11) Previous enrolment into the current study (12) Enrolment of the investigator, his/her family members, employees and other dependent persons

The exclusion criteria for the participants in the control group of healthy participants are:

1. Age younger than 6 and older than 65 years' old
2. Diagnosis of ADHD or other mental disorders
3. IQ-score lower than 80 points according to (WAIS-IV; Wechsler, 2008) and for children and adolescents according to (WISC-IV; Wechsler, 2003)
4. No written consent from participants and from the legal guardians of minors involved (for participants under 14 years old)
5. FMRI exclusion: claustrophobia, Pregnancy known or suspected, metallic implants in their bodies (e.g: pacemakers, aneurism clips, metal Prosthetic, cochlear implant)
6. In case of suicidal risk, the participant is encouraged to consult the medical staff.
7. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
8. Previous enrolment into the current study
9. Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-02-20 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
ADHD symptoms for adults | Change between two time points from baseline T1 to six week later T2 after cognitive training is assessed. Follow up is assessed at 3 months T3 and 6 months T4
  The Conners' Adult ADHD Rating Scales (CAARS) higher values represent worse outcome The Conners' Adult ADHD Rating Scales (CAARS) is used to assess ADHD symptoms among adults (Conners et al., 1999) depending on the DSM-IV-TR (APA, 2000). This short version includes 26 items and 4 possible ratings from from 0 (not at all) to 3 (very much). This scale comprises four factors: (1) inattention, memory problems, (2) hyperactivity, restlessness, (3) impulsivity, emotional lability, (4) problems with self-concept and one ADHD index. score are summed. Range 0 to 100.
ADHD symptoms for children | Change between two time points from baseline T1 to six week later T2 after cognitive training is assessed. Follow up is assessed at 3 months T3 and 6 months T4
  The Conners Scale, 3rd edition higher values represent a worse outcome Questionnaire is rated by the legal guardian. This questionnaire assesses ADHD symptoms.Score are summed. Score range 0 to 100.

SECONDARY OUTCOMES:
Impulsivity | Change between two time points from baseline T1 to six week later T2 after cognitive training is assessed. Follow up is assessed at 3 months T3 and 6 months T4
  The Impulsivity Behavior Scale (UPPS) higher values represent a worse outcome. score are summed short version contains 20 items measuring the following five dimensions of impulsivity: positive urgency, negative urgency, lack of perseverance, lack of premeditation and sensation seeking. This scale is based on Cyder and Smith (2007) and Whiteside and Lynam (2001) theory of impulsivity. Range 0 to 50.
executive function | Change between two time points from baseline T1 to six week later T2 after cognitive training is assessed. Follow up is assessed at 3 months T3 and 6 months T4
  The Behavior Rating Inventory of Executive Function higher values represent a worse outcome Score are summed. This questionnaire measures executive functionning in everyday life. The BRIEF includes 75 questions and eight sub-domains: Inhibit Shift, Emotional Control, Initiate, Working Memory, Plan/Organize, Organization of Materials and Monitor. Score range 0 to 100
Reward | Change between two time points from baseline T1 to six week later T2 after cognitive training is assessed. Follow up is assessed at 3 months T3 and 6 months T4
  Subjects will perform a reward under stress task adapted from the spatial delayed response task from (Glahn et al., 2002) measure reward (Martin-Soelch, C., et al.,2009: Gaillac et al., 2016). Reaction time is calculated.
  The sensitivity to Punishment and Sensitivity to Reward questionnaire for Children, adolescents (SPSRQ-C) (Colder and O'Connor 2004) and adults (SPSRQ, Torrubia, Ávila, Moltó, & Caseras, 2001) are used. These questionnaires are based on Gray's reinforcement sensitivity theory of personality (1981, 1987, 2000). Reward task higher values represent a better outcome. Score range 0 to 110.
Reward | Change between two time points from baseline T1 to six week later T2 after cognitive training is assessed. Follow up is assessed at 3 months T3 and 6 months T4
  The sensitivity to Punishment and Sensitivity to Reward questionnaire for Children, adolescents (SPSRQ-C) (Colder and O'Connor 2004) and adults (SPSRQ, Torrubia, Ávila, Moltó, & Caseras, 2001) are used. These questionnaires are based on Gray's reinforcement sensitivity theory of personality (1981, 1987, 2000). Reward task higher values represent a better outcome. Score range 0 to 110.
Memory | Change between two time points from baseline T1 to six week later T2 after cognitive training is assessed. Follow up is assessed at 3 months T3 and 6 months T4 training 4. Six months after cognitive training
  WISC-IV higher values represent a better outcome. The Wechsler Intelligence Scale for Children-Fourth Edition (WISC-IV, Wechsler, 2003) Score are standardized from 0 to 20 for subtest and summed from 0 to 150.
  The Wechsler Intelligence Scale for Children-Fourth Edition (WISC-IV, Wechsler, 2003) and the Weschler adult intelligent scale measure verbal memory. Score are standardized from 0 to 20 for subtest and summed from 0 to 150.
Memory | Change between two time points from baseline T1 to six week later T2 after cognitive training is assessed. Follow up is assessed at 3 months T3 and 6 months T4 training 4. Six months after cognitive training
  WAIS-IV higher values represent a better outcome .the Weschler adult intelligent scale to (WAIS-IV; Wechsler, 2008). Score are standardized from 0 to 20 for subtest and summed from 0 to 150.
  The Wechsler Intelligence Scale for Children-Fourth Edition (WISC-IV, Wechsler, 2003) and the Weschler adult intelligent scale measure verbal memory. Score are standardized from 0 to 20 for subtest and summed from 0 to 150.
Neural activity | Change between two time points from baseline T1 to six week later T2 after cognitive training is assessed. Follow up is assessed at 3 months T3 and 6 months T4
  The fMRI measure include. Resting-state functional MRI.Task-free. Subjects are instructed to just lie quietly in the scanner and to think of nothing in particular and let their mind wander.- binding potential (ΔBP) is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Amélie Dentz, Ph.D, Principal Investigator — University of Fribourg; Martin Soelch Chantal, PR, Principal Investigator — University of Fribourg
Locations (1):
- Dentz Amélie, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spencer-Smith M, Klingberg T. Correction: Benefits of a Working Memory Training Program for Inattention in Daily Life: A Systematic Review and Meta-Analysis. PLoS One. 2016 Nov 22;11(11):e0167373. doi: 10.1371/journal.pone.0167373. eCollection 2016. PMID 27875585
- [Result] Gathercole SE. Commentary: Working memory training and ADHD - where does its potential lie? Reflections on Chacko et al. (2014). J Child Psychol Psychiatry. 2014 Mar;55(3):256-7. doi: 10.1111/jcpp.12196. Epub 2014 Jan 20. PMID 24438534